CLINICAL TRIAL: NCT01660763
Title: P3 - A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of the Sufentanil NanoTab® PCA System/15 mcg (Zalviso™) for the Treatment of Post-Operative Pain in Patients After Knee or Hip Replacement Surgery
Brief Title: Efficacy and Safety Trial to Evaluate the Sufentanil NanoTab® PCA System/15 mcg (Zalviso™) for Post-Operative Pain in Patients After Knee or Hip Replacement Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IAP311
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sufentanil NanoTab PCA System/15 mcg (Experimental)
  Interventions: Drug: Sufentanil NanoTab PCA System/15 mcg
- Placebo Sufentanil NanoTab PCA System (Placebo Comparator)
  Interventions: Drug: Placebo Sufentanil NanoTab PCA System

INTERVENTIONS:
Drug: Sufentanil NanoTab PCA System/15 mcg — 15 mcg Sufentanil NanoTab dosed sublingually every 20 minutes as needed for pain for at least 48 hours. Patients may elect to remain in study for up to 72 hours.
  Other Names: sufentanil sublingual microtablet system; Zalviso™
  Arms: Sufentanil NanoTab PCA System/15 mcg
Drug: Placebo Sufentanil NanoTab PCA System — Placebo NanoTab dosed sublingually every 20 minutes as needed for pain for at least 48 hours. Patients may elect to remain in study for up to 72 hours.
  Arms: Placebo Sufentanil NanoTab PCA System

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the Sufentanil NanoTab PCA System/15 mcg to the Placebo Sufentanil NanoTab PCA System for the management of acute moderate to severe post-operative pain after total unilateral knee or total unilateral hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 18 years of age or older
* Patients who are scheduled for an elective cemented or uncemented total unilateral knee replacement or total unilateral hip replacement, under general or spinal anesthesia that does not include use of an intrathecal opioid
* Post-surgical patients who have been admitted to the PACU and are expected to remain hospitalized and to have acute post-operative pain requiring parenteral opioids for at least 48 hours after surgery

Exclusion Criteria:

* Patients who have undergone a replacement of the same knee or hip
* Patients who have taken an opioid for more than 30 consecutive days, at a daily dose of more than 15 mg of morphine (or equivalent), within the past 3 months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet)
* Patients with an allergy or hypersensitivity to opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Palmer, M.D., PhD, Study Director — Chief Medical Officer, AcelRx Pharmaceuticals, Inc.
Locations (1):
- Deidre Stonestreet, Damascus, Maryland, United States

REFERENCES:
- [Background] Jove M, Griffin DW, Minkowitz HS, Ben-David B, Evashenk MA, Palmer PP. Sufentanil Sublingual Tablet System for the Management of Postoperative Pain after Knee or Hip Arthroplasty: A Randomized, Placebo-controlled Study. Anesthesiology. 2015 Aug;123(2):434-43. doi: 10.1097/ALN.0000000000000746. PMID 26079801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period of 9 months - August 2012 through April 2013
Pre-assignment Details: Patients were excluded per protocol exclusion criteria at Screening as well as post surgery for certain conditions including the following:
  1. Patients who were not awake or stable
  2. Patients with arterial oxygen saturation that couldn't be maintained at 95% or greater
  3. Patients with uncontrollable vomiting
Groups:
- Sufentanil NanoTab PCA System/15 mcg: Sufentanil NanoTab PCA System/15 mcg : 15 mcg Sufentanil NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours and up to 72 hours
- Placebo Sufentanil NanoTab PCA System: Placebo Sufentanil NanoTab PCA System : Placebo NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours and up to 72 hours
Period: Overall Study
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System
Started | 315 | 104
Completed | 215 | 43
Not Completed | 100 | 61
Not completed — Lack of Efficacy | 45 | 50
Not completed — Adverse Event | 22 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Patient ready for early discharge | 28 | 4

BASELINE CHARACTERISTICS:
Groups:
- Sufentanil NanoTab PCA System/15 mcg: Sufentanil NanoTab PCA System/15 mcg : 15 mcg Sufentanil NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours. Patient may elect to remain in study for up to 72 hours
- Placebo Sufentanil NanoTab PCA System: Placebo Sufentanil NanoTab PCA System : Placebo NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours. Patient may elect to remain in study for up to 72 hours
- Total: Total of all reporting groups
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System | Total
Number analyzed (Participants) | 315 | 104 | 419
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 50 | 179
  >=65 years | 186 | 54 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.8) | 65.0 (10.5) | 66.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 66 | 254
  Male | 127 | 38 | 165
Region of Enrollment [Number; unit: participants]
  United States | 315 | 104 | 419

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 48-hour Study Period (SPID48).
Description: SPID-48 is the sum of the pain intensity difference (PID) over the 48 hour time period. A pain intensity score of 0 (no pain) to 10 (worse possible pain) is obtained before starting the study and throughout the 48 time period. The pain score at each assessment time is subtracted from the baseline pain score to provide the total sum score or SPID-48. A higher SPID-48 is better and indicates a reduction in pain intensity compared to the baseline score. Range of SPID48 scores were -239 to 417.
  Time-weighted SPID48 = ∑ [T(i) - T(i-1)] x PID(i), where T(0) = Time 0 (baseline), T(i) is the scheduled or unscheduled assessment time, and PID(i) is the PID score at time i for i=0 to 48 hours
Time Frame: 48 hours
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Sufentanil NanoTab PCA System/15 mcg: Sufentanil NanoTab PCA System/15 mcg : 15 mcg Sufentanil NanoTab dosed sublingually every 20 minutes as needed for pain for up to 48 hours. Patients may elect to remain in study for up to 72 hours.
- Placebo Sufentanil NanoTab PCA System: Placebo Sufentanil NanoTab PCA System/15 mcg : Placebo NanoTab dosed sublingually every 20 minutes as needed for pain for up to 48 hours. Patients may elect to remain in study for up to 72 hours.
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System
Number analyzed (Participants) | 315 | 104
Units on a scale | 76.24 (7.02) | -11.35 (10.55)
Statistical Analysis 1: Comparison: Sufentanil NanoTab PCA System/15 mcg vs Placebo Sufentanil NanoTab PCA System; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 87.59, 95% CI 2-sided [66.20 to 108.98], Standard Error of Mean 10.88

ADVERSE EVENTS:
Time Frame: AEs were collected from time of first study drug dose taken through 12 hours after last study drug dose taken.
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System
Serious Adverse Events (participants affected / at risk) | 8/315 | 4/104
Other Adverse Events (participants affected / at risk) | 171/315 | 35/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab PCA System/15 mcg (N=315) | Placebo Sufentanil NanoTab PCA System (N=104)
Acute Renal Failure (Renal and urinary disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0
Coagulopathy (Investigations) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Epididymitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fecal Infection (Gastrointestinal disorders) | 0 | 1 — Faecaloma
Hypoxia (Investigations) | 1 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Aspiration Pneumonia
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab PCA System/15 mcg (N=315) | Placebo Sufentanil NanoTab PCA System (N=104)
Confusional State (Psychiatric disorders) | 8 | 1
Constipation (Gastrointestinal disorders) | 15 | 1 — All AEs in this table were assessed by the PI as possibly or probably related to study drug
Dizziness (Nervous system disorders) | 16 | 1
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Headache (Nervous system disorders) | 13 | 6
Hypotension (Vascular disorders) | 12 | 2
Insomnia (Psychiatric disorders) | 13 | 3
Nausea (Gastrointestinal disorders) | 110 | 23
Orthostatic Hypotension (Vascular disorders) | 4 | 2
Oxygen Saturation Decreased (Investigations) | 22 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 0
Pyrexia (General disorders) | 4 | 2
Sedation (Nervous system disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 34 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days